CLINICAL TRIAL: NCT05999773
Title: Potential Role of Sodium Glucose Cotransporter 2 Inhibitors in the Treatment of Ascites in Cirrhotic Patients
Brief Title: SGLT-2 Inhibitors in the Treatment of Ascites
Status: Recruiting | Type: Observational
Sponsor: University of Palermo (Other)
Collaborators: Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello (Other)
Responsible Party: Principal Investigator, Aurelio Seidita, Medical Doctor, University of Palermo
Other Study IDs: ASLG01
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Ascites Hepatic; Cirrhosis, Liver; Diabete Type 2
Keywords: Ascites; Liver Cirrhosis; Diabete Type 2; Sodium Glucose Cotransporter 2 (SGLT-2) Inhibitors; Glyphozines
MeSH Terms: conditions — Liver Cirrhosis; Diabetes Mellitus, Type 2; Ascites | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SGLT-2i Group: Patients diagnosed with Child-Turcotte-Pugh A6-B9 class Hepatic Cirrhosis (moderately impaired liver function) and type 2 Diabetes Mellitus assigned to start SGLT-2 inhibitors intake, according diabetology indications, in addition to standard medical therapy for 6 months.
  Interventions: Drug: SGLT2 inhibitor
- Standard Therapy Group: Patients diagnosed with Child-Turcotte-Pugh A6-B9 class Hepatic Cirrhosis (moderately impaired liver function) and type 2 Diabetes Mellitus assigned to continue standard medical therapy, according diabetology indications, for 6 months.

INTERVENTIONS:
Drug: SGLT2 inhibitor — Start of SGLT-2 inhibitors to treat diabetes according diabetology indications.
  Groups: SGLT-2i Group

SUMMARY:
The goal of this observational study is to test the efficacy of glyphozines (SGLT-2 inhibitors) in the control of ascites in patients with liver cirrhosis in class A6-B9, according to the Child-Pugh classification, and type 2 diabetes mellitus. The investigators will compare patients belonging to the intervention group (A), who will be given SGLT-2 inhibitors according to diabetology indications in addition to standard medical therapy for 6, with patients of the control group (B), who will, instead, continue with the standard medical therapy for 6 months. Standard medical therapy will include dietary sodium restriction, treatment with diuretics (furosemide and spironolactone), hypoglycemic therapy (metformin, insulin, or both) and other supportive care.

The main questions aims of this study are:

1. Compare the efficacy and safety of a therapeutic approach based on the administration of SGLT-2 inhibitors in addition to optimal medical therapy (MRA and loop diuretic) compared to traditional diuretic therapy only, in cirrhotic patients with saline retention and diabetes.
2. Demonstrate better control of the glycemic profile in cirrhotic diabetic patients using SGLT-2 inhibitors.

DETAILED DESCRIPTION:
Background The occurrence of ascites and saline retention is the most common complication in patients affected by liver cirrhosis and it is associated with poor prognosis.

It is well-known that in liver cirrhosis the underlying pathogenetic events responsible of ascites are portal hypertension and splanchnic vasodilation. These mechanisms reduce the effective circulating blood volume, triggering counter-regulatory systems such as the sympathetic nervous system (SNS) and the renin-angiotensin-aldosterone system (RAAS), that leading to renal sodium and water retention.

Therefore, considering pathogenetic knowledge, the cornerstones of ascites treatment are sodium restriction and drugs such as mineralocorticoid receptor antagonists (MRA) and loop diuretics, reserving more invasive techniques, like paracentesis with administration of human albumin, for more severe patients with grade 3 ascites unresponsive to diuretics. However, even though diuretics have proven to be among the most efficient drugs in controlling ascites, patients with liver cirrhosis and ascites treated with diuretics develop adverse drug reactions in 20-40% of cases.

One of the most common comorbidities of liver cirrhosis is type-2 diabetes mellitus (DM2), which affects approximately one-third of cirrhotic patients. The connection between liver cirrhosis and DM2 is complex. DM2 can be a secondary effect or, conversely, a casual factor of liver dysfunction.

Sodium glucose cotransporter 2 inhibitors (SGLT-2i) are a relatively new class of drugs for the management of type-2 diabetes mellitus. They inhibit the reabsorption of sodium and glucose in the proximal convoluted tubule of the nephron, leading to a significant natriuresis and have proven to be effective and safe drugs for the control of the glycemic profile in patients with liver dysfunction.

In recently published case reports, SGLT-2i have also proven to be safe and effective in controlling the glycemic profile in patients with liver dysfunction. In these patients, in addition to better control the glycemic profile, they led to saline retention improvement and to weight loss, without inducing encephalopathy or acute kidney injury. Other studies have hypothesized that, similarly to the previously demonstrated beneficial effect of glyphozines in patients with acute heart failure, SGLT-2i may also lead to the improvement of complicated liver cirrhosis acting as "neuromodulators", suppressing the RAAS axis and inducing better mobilization of ascites and reduction of saline retention.

Currently, there are no randomized controlled trials supporting these evidences.

In this observational study the investigators intend to evaluate the efficacy and safety of SGLT-2i in cirrhotic and diabetic patients with saline retention.

Aims

* Comparing the efficacy and safety of a therapeutic approach based on the administration of SGLT-2i in addition to optimal medical therapy (MRA and loop diuretic) compared to traditional diuretic therapy only, in cirrhotic patients with saline retention and diabetes.
* Demonstrating better control of the glycemic profile in cirrhotic diabetic patients using SGLT-2i.

Sample and study design Our study will be a clinical, prospective, observational multicenter study. The investigators will enroll subjects with complicated liver cirrhosis and type II diabetes mellitus consecutively, in two centers: Internal Medicine Unit of the "Policlinico Paolo Giaccone", University Hospital of Palermo, Italy and Internal Medicine Unit of the "Ospedali Riuniti Villa Sofia- Cervello" Hospital of Palermo, Italy.

Sample size The sample size is difficult to determine as there are no studies that have evaluated the efficacy of SGLT-2i treatment in addition to diuretic therapy in the patient with liver cirrhosis and saline retention. To date, there are only a few case reports in the literature that have demonstrated its effectiveness. Considering the prospective and pilot nature of this study the investigators decided to enroll at least 40 patients.

Study design and outcome evaluation Our project has been approved by the ethics committee of the University Hospital of Palermo.

Patients enrolled on the basis of the inclusion and exclusion criteria and who agreed to enter the study, after signing the informed consent, will be assigned to intervention group (group A) or control group (group B).

Patients belonging to the intervention group (A) will be given SGLT-2 inhibitors, according diabetology indications, in addition to standard medical therapy for 6 months; the patients of the control group (B) will instead continue with the only standard medical therapy for 6 months, according diabetology indications.

Standard medical therapy will include dietary sodium restriction, treatment with diuretics (furosemide and spironolactone), hypoglycemic therapy (metformin, insulin, or both) and other supportive care. Patients taking non-selective beta-blockers will continue to do.

Patients in group A and group B will be evaluated for specific clinical and laboratory parameters before the start of the study (T0) and they will subsequently be evaluated again at 4 weeks, 3 months and 6 months (T1, T2, T3).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Patients diagnosed with Child-Turcotte-Pugh A6-B class Hepatic Cirrhosis (moderately impaired liver function)
* Patients diagnosed with Hepatic Cirrhosis of viral etiology (if previous hepatitis C virus (HCV) infection they must be in Sustained Virological Response (SVR); if previous hepatitis B virus (HBV) infection they must have undetectable viral genome)
* Patients diagnosed with hepatic cirrhosis of metabolic etiology
* Patients diagnosed with liver cirrhosis of alcoholic etiology (non active potus)
* Patients with grade 1 ascites: ascites detectable only ultrasound that can be fully mobilized or controlled with diuretic therapy associated with or without moderate dietary sodium restriction
* Grade 2 ascites: ascites that leads to a moderate abdominal distension and that recurs on at least 3 occasions within a 12-month period despite sodium restriction and adequate diuretic therapy (23)
* Patients diagnosed with type II diabetes mellitus defined according to 2022 American Diabetes Association (ADA) guidelines.

Exclusion Criteria:

* Inability to obtain informed consent
* Ascites of non-cirrhotic origin
* Patients diagnosed with heart failure Heart (NYHA) class => 2
* Patients diagnosed with acute renal failure
* Patients diagnosed with chronic renal failure and glomerular filtration rate (eGFR) below 25ml/min
* Patients with hepatocellular carcinoma (diagnosed according to the Barcelona criteria) or other active tumors (25)
* Grade 3 ascites: ascites that causes marked distention of the abdomen and that cannot be mobilized or whose early recurrence (i.e. after large volume paracentesis) cannot be satisfactorily prevented by medical therapy
* Patients diagnosed with acute Spontaneous Bacterial Peritonitis (26)
* Patients diagnosed with severe hepatic encephalopathy
* Patients diagnosed with autoimmune diseases on active steroid treatment
* Patients diagnosed with liver cirrhosis due to storage diseases
* Patients diagnosed with cirrhosis of the liver due to enzyme deficiency
* Patients diagnosed with complete portal thrombosis
* Patients with active sepsis
* Pregnant or breastfeeding women
* Patients who use drugs
* Patients with active alcohol consumption

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll subjects with complicated liver cirrhosis and type II diabetes mellitus consecutively, in two centers: Internal Medicine Unit of the "Policlinico Paolo Giaccone", University Hospital of Palermo, Italy and Internal Medicine Unit of the "Ospedali Riuniti Villa Sofia- Cervello" Hospital of Palermo, Italy.
  Patients will be assigned to intervention or control group according diabetology indications to start SGLT-2 inhibitors.
  Patients included in the two study groups will be sex, age and race matched.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ascites control | Day 0, 4 weeks, 3 months, 6 months
  Ascites control, defined in terms of:
  * Optimal control, in case of total disappearance of the ascites
  * Reduction of the grade of ascites from grade 2 to grade 1 (i.e. ascites that is clinically undetectable, which does not determine abdominal distension and detectable only by ultrasound).
  * Absence of response, in case of persistence of ascites of the same degree.
Glycemic control | Day 0, 4 weeks, 3 months, 6 months
  Reduction of glycosylated hemoglobin (HbA1C) levels from baseline to the end of the study, defined as:
  * Optimal control: HbA1C below 6.5%
  * Good control: HbA1C between 6.5% and 6.9%
  * Inadequate control: HbA1C between 7.0% and 8%
  * Poor control: HbA1C above 8.0%
SGLT-2 inhibitors related adverse events | Day 0, 4 weeks, 3 months, 6 months
  Appearance of any adverse effect related to the intake of an SGLT-2 inhibitor, classified as follows:
  * None: no adverse effects
  * Minimal: adverse effect which does not significantly compromise the patient's state of health and which allows the continuation of the therapy
  * Moderate: adverse effect which significantly compromises the patient's state of health and which does not allow the continuation of the therapy, managed in an outpatient setting.
  * Severe: adverse effect which significantly compromises the patient's state of health and which does not allow the continuation of the therapy, managed in an inpatient setting.
  * Life-threatening: adverse effect that puts the patient's life in danger and which requires the immediate interruption of therapy and hospitalization.

SECONDARY OUTCOMES:
Fasting glucose control | Day 0, 4 weeks, 3 months, 6 months
  Fasting blood glucose will be evaluated by finger stick glucose auto measurement after overnight fasting in the 5 days preceding the outpatient visit, and will be classified as:
  - Good fasting glucose control: average of three consecutive fasting blood glucose measurement between 80-130 mg/dl.
  Poor glycemic control: average blood glucose measurements of three consecutive fasting blood glucose measurement >130 or <70 mg/dl
Weight loss | Day 0, 4 weeks, 3 months, 6 months
  Weight reduction will be assessed by weight measurements at day 0, at 4 weeks, 3 months and 6 months, and will be classified as:
  * Optimal: weight loss >= 5 kg
  * Good: 5 Kg< weight loss =< 2.5 Kg
  * Poor: 2.5 Kg< weight loss < 0 Kg
  * Gain: any value of weight gain
24-hour diuresis | Day 0, 4 weeks, 3 months, 6 months
  24-hours diuresis will be assessed at day 0, at 4 weeks, 3 months and 6 months and will be classified as:
  * None: no change in 24- hours urinary volume
  * Decrease: significant (p<0.05) reduction of 24- hours urinary volume
  * Increase: significant (p<0.05) increase of 24- hours urinary volume
Sodium excretion in the urine | From day 0 to day 180
  Fraction of sodium excretion will be evaluated on 24-hours diuresis at day 0, at 4 weeks, 3 months and 6 months and will be classified as:
  * None: no change in 24- hours sodium excretion
  * Decrease: significant (p<0.05) reduction of 24- hours sodium excretion
  * Increase: significant (p<0.05) increase of 24- hours sodium excretion
Natremia | Day 0, 4 weeks, 3 months, 6 months
  Natremia will be evaluated on plasma samples at day 0, at 4 weeks, 3 months and 6 months and will be classified as:
  * None: no change in natremia
  * Decrease: significant (p<0.05) reduction of natremia
  * Increase: significant (p<0.05) increase of natremia
Mean arterial pressure | Day 0, 4 weeks, 3 months, 6 months
  Mean arterial pressure will be evaluated according international guidelines of blood pressure assessment at day 0, at 4 weeks, 3 months and 6 months and will be classified as:
  * None: no change in mean arterial pressure
  * Decrease: significant (p<0.05) reduction of mean arterial pressure
  * Increase: significant (p<0.05) increase of mean arterial pressure
Glomerular filtration rate | Day 0, 4 weeks, 3 months, 6 months
  Glomerular filtration rate will be evaluated according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) measurement at day 0, at 4 weeks, 3 months and 6 months and will be classified as:
  * None: no change in glomerular filtration rate
  * Decrease: significant (p<0.05) reduction of glomerular filtration rate
  * Increase: significant (p<0.05) increase of glomerular filtration rate
Child-Turcotte-Pugh (CTP) score | Day 0, 4 weeks, 3 months, 6 months
  CTP score will be evaluated at day 0, at 4 weeks, 3 months and 6 months and will be classified as:
  * None: no change in glomerular filtration rate
  * Reduction: decrease of at least 1 point in the CTP score
  * Increase: increase of at least 1 point in the CTP score
Survival | 6 months
  Overall patient's survival will be evaluated after 6 months from the study enrollment
Loop diuretics posology | Day 0, 4 weeks, 3 months, 6 months
  Loop diuretics posology (mg/die) will be evaluated at day 0, at 4 weeks, 3 months and 6 months and will be classified as:
  * None: no change in loop diuretics posology to control ascites
  * Reduction: decrease of loop diuretics posology to control ascites
  * Increase: increase of loop diuretics posology to control ascites
Mineralocorticoid receptor antagonists posology | Day 0, 4 weeks, 3 months, 6 months
  Mineralocorticoid receptor antagonists diuretics posology (mg/die) will be evaluated at day 0, at 4 weeks, 3 months and 6 months and will be classified as:
  * None: no change in mineralocorticoid receptor antagonists posology to control ascites
  * Reduction: decrease of mineralocorticoid receptor antagonists posology to control ascites
  * Increase: increase of mineralocorticoid receptor antagonists posology to control ascites
Metformin posology | Day 0, 4 weeks, 3 months, 6 months
  Metformin (only in patients taking metformin) posology (mg/die) will be evaluated at day 0, at 4 weeks, 3 months and 6 months and will be classified as:
  * None: no change in metformin posology to control ascites
  * Reduction: decrease of metformin posology to control ascites
  * Increase: increase of metformin posology to control ascites
Insulin bolus posology | Day 0, 4 weeks, 3 months, 6 months
  Insulin bolus (only in patients taking insulin) posology (mg/die) will be evaluated at day 0, at 4 weeks, 3 months and 6 months and will be classified as:
  * None: no change in insulin bolus posology to control ascites
  * Reduction: decrease of insulin bolus posology to control ascites
  * Increase: increase of insulin bolus posology to control ascites
Insulin basal posology | Day 0, 4 weeks, 3 months, 6 months
  Insulin basal (only in patients taking insulin) posology (mg/die) will be evaluated at day 0, at 4 weeks, 3 months and 6 months and will be classified as:
  * None: no change in insulin basal posology to control ascites
  * Reduction: decrease of insulin basal posology to control ascites
  * Increase: increase of insulin basal posology to control ascites
Adverse events classification | 4 weeks, 3 months, 6 months
  Putative adverse events related to SGLT-2 inhibitors intake will be classified as:
  * Allergy: appearance of any allergic manifestation including: skin rash, itching, erythema, urticaria, angioedema, anaphylaxis, anaphylactic shock
  * Infectious diseases: Occurrence of any of the following conditions: Vulvovaginal candidiasis, balanitis or balanoposthitisb, urinary tract infection (including pyelonephritis and urosepsis)
  * Metabolism disorders: hypoglycemia, dehydration, diabetic ketoacidosis, dyslipidemia, hyperkalaemia, hyperphosphoraemia
  * Nervous system disorders: postural dizziness, syncope
  * Vascular disorders: hypotension, orthostatic hypotension
  * Gastrointestinal disorders: constipation, thirst, nausea
  * Musculoskeletal system disorders: bone fracture
  * Renal and urinary disorders: polyuria, pollakiuria, renal insufficiency (mainly in the context of hypovolemia)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Giannitrapani, MD, Principal Investigator — University of Palermo
Locations (2):
- Italy (2):
  - Internal Medicine Unit, V. Cervello Hospital, Palermo, Italy
  - Department of Internal Medicine, University Hospital of Palermo, Palermo, Palermo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bernardi M, Moreau R, Angeli P, Schnabl B, Arroyo V. Mechanisms of decompensation and organ failure in cirrhosis: From peripheral arterial vasodilation to systemic inflammation hypothesis. J Hepatol. 2015 Nov;63(5):1272-84. doi: 10.1016/j.jhep.2015.07.004. Epub 2015 Jul 17. PMID 26192220
- [Background] Angeli P, Gatta A, Caregaro L, Menon F, Sacerdoti D, Merkel C, Rondana M, de Toni R, Ruol A. Tubular site of renal sodium retention in ascitic liver cirrhosis evaluated by lithium clearance. Eur J Clin Invest. 1990 Feb;20(1):111-7. doi: 10.1111/j.1365-2362.1990.tb01800.x. PMID 2108033
- [Background] Santos J, Planas R, Pardo A, Durandez R, Cabre E, Morillas RM, Granada ML, Jimenez JA, Quintero E, Gassull MA. Spironolactone alone or in combination with furosemide in the treatment of moderate ascites in nonazotemic cirrhosis. A randomized comparative study of efficacy and safety. J Hepatol. 2003 Aug;39(2):187-92. doi: 10.1016/s0168-8278(03)00188-0. PMID 12873814
- [Background] Garcia-Compean D, Gonzalez-Gonzalez JA, Lavalle-Gonzalez FJ, Gonzalez-Moreno EI, Maldonado-Garza HJ, Villarreal-Perez JZ. The treatment of diabetes mellitus of patients with chronic liver disease. Ann Hepatol. 2015 Nov-Dec;14(6):780-8. doi: 10.5604/16652681.1171746. PMID 26436350
- [Background] Kasichayanula S, Liu X, Zhang W, Pfister M, LaCreta FP, Boulton DW. Influence of hepatic impairment on the pharmacokinetics and safety profile of dapagliflozin: an open-label, parallel-group, single-dose study. Clin Ther. 2011 Nov;33(11):1798-808. doi: 10.1016/j.clinthera.2011.09.011. Epub 2011 Oct 26. PMID 22030444
- [Background] Montalvo-Gordon I, Chi-Cervera LA, Garcia-Tsao G. Sodium-Glucose Cotransporter 2 Inhibitors Ameliorate Ascites and Peripheral Edema in Patients With Cirrhosis and Diabetes. Hepatology. 2020 Nov;72(5):1880-1882. doi: 10.1002/hep.31270. No abstract available. PMID 32294260
- [Background] Kalambokis GN, Tsiakas I, Filippas-Ntekuan S, Christaki M, Despotis G, Milionis H. Empagliflozin Eliminates Refractory Ascites and Hepatic Hydrothorax in a Patient With Primary Biliary Cirrhosis. Am J Gastroenterol. 2021 Mar 1;116(3):618-619. doi: 10.14309/ajg.0000000000000995. No abstract available. PMID 33027081
- [Background] Saffo S, Taddei T. SGLT2 inhibitors and cirrhosis: A unique perspective on the comanagement of diabetes mellitus and ascites. Clin Liver Dis (Hoboken). 2018 Jul 26;11(6):141-144. doi: 10.1002/cld.714. eCollection 2018 Jun. No abstract available. PMID 30992805
- [Background] Gao Y, Wei L, Zhang DD, Chen Y, Hou B. SGLT2 Inhibitors: A New Dawn for Recurrent/Refractory Cirrhotic Ascites. J Clin Transl Hepatol. 2021 Dec 28;9(6):795-797. doi: 10.14218/JCTH.2021.00418. Epub 2021 Nov 26. No abstract available. PMID 34966642